CLINICAL TRIAL: NCT06966479
Title: A Long-Term Extension Study to Evaluate Safety and Efficacy of Verekitug (UPB-101) in Adult Participants With Severe Asthma Who Completed the VALIANT Trial
Brief Title: A Long-Term Safety and Efficacy Study of Verekitug (UPB-101) in Adult Participants With Severe Asthma (VALOUR)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Upstream Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPB-CP-05; 2024-519469-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-09; First posted 2025-05-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Severe Asthma
Keywords: UPB-101; Verekitug; TSLP receptor; monoclonal antibody; VALIANT; VALOUR; Respiratory Tract Diseases; Bronchial Diseases; Asthma; Lung Diseases; Uncontrolled Asthma
MeSH Terms: conditions — Asthma; Respiratory Tract Diseases; Bronchial Diseases; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Verekitug 100 mg Q12W and Placebo (Experimental): Participants will receive 0.5 mL of verekitug (100 mg) and 2.0 mL of matching placebo, subcutaneous (SC) injections, every 12 weeks (Q12W) for up to 48 weeks.
  Interventions: Drug: Verekitug; Drug: Placebo
- Verekitug 400 mg Q24W and Placebo (Experimental): Participants will receive 2.0 mL of verekitug (400 mg) and 0.5 mL of matching placebo, SC injections, at Weeks 24 and 48 visits. Participants will also receive 2.0 mL and 0.5 mL of placebo subcutaneously in two separate injections at Weeks 12 and 36 visits.
  Interventions: Drug: Verekitug; Drug: Placebo

INTERVENTIONS:
Drug: Verekitug — Verekitug subcutaneous injection.
  Other Names: UPB-101
Drug: Placebo — Verekitug matching placebo.

SUMMARY:
The primary purpose of this study is to evaluate the long-term safety and efficacy of verekitug (UPB-101) in participants who complete the VALIANT study (NCT06196879).

ELIGIBILITY:
Inclusion Criteria:

1. Completion of the VALIANT study (UPB-CP-04 [NCT06196879]) per protocol.
2. Participant has signed, dated, and received a copy of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent form (ICF) for the LTE study.
3. Contraceptive use by participants must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Abnormal medical history, physical finding, or safety finding that in the opinion of the Investigator may obscure the study data or interfere with the participant's safety.
2. Any clinical laboratory test result outside of the reference ranges considered by the Investigator as clinically significant and that may obscure the study data or interfere with the participant's safety.
3. Participant with a history or evidence of a clinically significant pulmonary condition (other than asthma), including significant restrictive findings on pulmonary function testing, chronic bronchitis, emphysema, bronchiectasis, pulmonary fibrosis, or any other related condition that may obscure the study data (e.g., gastroesophageal reflux and vocal cord paralysis/dysfunction).
4. Pregnant or breastfeeding or planning to become pregnant or breastfeed during the study or unwilling to use adequate birth control, if of reproductive potential and sexually active.
5. Participants with significant protocol deviations in VALIANT, assessed at the discretion of the Sponsor.
6. Participant is unreliable, incapable of adhering to the protocol and visit schedule according to the judgment of the Investigator or has any disorder that may compromise their ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From VALOUR baseline up to Week 64
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Annualized Asthma Exacerbation Rate (AAER) | From VALOUR baseline up to Week 60
  An asthma exacerbation is defined as a worsening of asthma that required treatment with systemic (oral or intravenous) corticosteroids for at least three consecutive days or a single depo-injectable dose of corticosteroids or an emergency room (ER) or urgent care visit that required systemic corticosteroids or an admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for greater than or equal to 24 hours.
Change from LTE Baseline in Forced Expiratory Volume in 1 Second (FEV1) | From VALOUR baseline to Week 60
  Spirometry will be performed pre-bronchodilator (BD) to measure lung function. FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Change from LTE Baseline in Fractional Exhaled Nitric Oxide (FeNO) | From VALOUR baseline up to Week 60
  Standardized single breath FeNO test is performed to evaluate airway inflammation.
Change from LTE Baseline in Asthma Control Questionnaire-6 (ACQ-6) | From VALOUR baseline to Week 60
  ACQ-6 is a participant-reported questionnaire to assess asthma control with 6 items assessing night-time waking, symptoms on waking, activity limitation, shortness of breath, wheeze, and rescue short-acting beta agonist use. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 score is the mean of the responses.

CONTACTS AND LOCATIONS:
Overall Officials: James C Lee, MD, Study Director — Upstream Bio
Locations (57):
- United States (24):
  - Kern Research, Inc., Bakersfield, California
  - California Medical Research Associates Inc., Northridge, California
  - Integrated Research of Inland Inc, Upland, California
  - Allianz Research Institute, Westminster, California
  - Phoenix Medical Research, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Health and Life Research Institute, LLC, Miami, Florida
  - Nouvelle Clinical Research, Miami, Florida
  - Edward Jenner Research Group, LLC, Plantation, Florida
  - R&B Medical Center, Tampa, Florida
  - Clinical Site Partners dba Flourish research, Winter Park, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Chesapeake Clinical Research Inc, White Marsh, Maryland
  - Pulmonary Research Institute of Southeast Michigan (PRISM), Farmington Hills, Michigan
  - AA MRC, Flint, Michigan
  - M3 Wake Research, Las Vegas, Nevada
  - Urban Health Plan INC, The Bronx, New York
  - Toledo Institute of Clinical Research Inc, Toledo, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Alina Clinical Trials, LLC, Dallas, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - California Medical Research Associates Inc., Houston, Texas
  - Metroplex Pulmonary and Sleep Center Drive, McKinney, Texas
  - DM Clinical Tomball, Tomball, Texas
- Argentina (2):
  - Instituto de Medicina Respiratoria, IMeR/ Instituto Médico DAMIC, Córdoba, Córdoba Province
  - Fundacion Scherbovsky, Mendoza, Mendoza Province
- Bulgaria (5):
  - MHAT "Rahila Angelova" Pernik, Pernik, Pernik
  - Ambulatory For Specialized Outpatient Medical Care - Individual Practice - Dr. Nikolay Evgeniev Ruse Ltd, Rousse, Ruse
  - Medical Center Excelsior (Todor Popov), Sofia, Sofia
  - MC Convex/DCC Convex, Sofia, Sofia
  - Medical Center New Rehabilitation Center EOOD, Stara Zagora, Stara Zagora
- Dynamic Drug Advancement, Ajax, Ontario, Canada
- Germany (3):
  - RCMS/Lungenpraxis Hohenzollerndamm, Berlin, Germany
  - POIS Sachsen GmbH, Leipzig, Germany
  - ME Clinical Respiratory Research Hamburg GmbH, Hamburg, Hamburg
- Japan (5):
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - Oji General Hospital, Hokkaido, Hokkaido
  - Osaka Habikino Medical Center, Osaka, Japan
  - Kishiwada City Hospital, Osaka, Japan
  - Fukuwa Clinic, Tokyo, Tokyo
- Poland (9):
  - ALL-MED Specjalistyczna Opieka Medyczna. Medyczny Instytut Badawczy Marek Jutel, Wroclaw, Dolnoslaskie Voivodeship
  - NZOZ J. Małolepszy i Partnerzy, Wroclaw, Dolnoslaskie Voivodeship
  - Centrum Medyczne "All-Med" Badania Kliniczne, Krakow, Malopolskie Voivodeship
  - ATOPIA Niepubliczny Zakład Opieki Zdrowotnej Poradnie Specjalistyczne, Krakow, Malopolskie Voivodeship
  - Małopolskie Centrum Alergologii Spółka z ograniczoną odpowiedzialnością, Krakow, Malopolskie Voivodeship
  - "Alergo-Med" Specjalistyczna Przychodnia Lekarska Spolka Z Ograniczona Odpowiedzialnoscia, Tarnów, Malopolskie Voivodeship
  - Prywatny Gabinet Lekarski Malgorzata Pawlukiewicz, Rzeszów, Podkarpackie Voivodeship
  - Centrum Medycyny Oddechowej, Mroz Spolka Jawna, Bialystok, Podlaskie Voivodeship
  - Ostrowieckie Centrum Medyczne spolka cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Allergy & Immunology Unit, UCT Lung Institute, Cape Town, Western Cape, South Africa
- South Korea (3):
  - Yeungnam University Hospital, Daegu, Republic of Korea
  - Chungbuk National University Hospital, Jungbuk, Republic of Korea
  - Asan Medical Center, Seoul, Republic of Korea
- Spain (2):
  - Pectus Respiratory Health, Barcelona, Catalonia
  - Hospital Gregorio Marañon, Madrid, Madrid
- United Kingdom (2):
  - Castle Hill Hospital, Hull University Teaching Hospitals NHS Trust, Cottingham, East Yorkshire
  - Gartnavel General Hospital (Glasgow Clinical Research Facility), Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No